CLINICAL TRIAL: NCT06907836
Title: Description of a Retrospective Cohort of Patients With Transthyretin Cardiac Amyloidosis (ATTR-CA) in Internal Medicine
Acronym: ATTR-CA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9302
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac Amyloidosis; Internal medicine
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2024, the prevalence of TTR cardiac amyloidosis is difficult to determine precisely. Indeed, the disease has long been underdiagnosed due to a lack of effective treatment and non-invasive diagnostic methods. The prevalence of ATTRwt is estimated at 155 to 191 cases per million person-years, with an incidence of 36 cases per million person-years. Both incidence and prevalence increase with age.

The most common presentation of TTR cardiac amyloidosis is heart failure with preserved ventricular ejection fraction (LVEF).

The natural history of TTR cardiac amyloidosis is progression to restrictive heart disease with all the complications described above.

The median time between diagnosis and the first cardiac symptoms was 39 months. Currently, the median survival in France is approximately 3.5 years, but survival appears to be improving, with a mortality rate of 73.5% at 30 months between 2002 and 2006, compared to 15% at 60 months between 2017 and 2022.

The number of patients diagnosed with TTR cardiac amyloidosis appears to be increasing. The overwhelming majority of available data concerns patients treated in cardiology. However, the issue of TTR cardiac amyloidosis concerns all specialists caring for patients with heart failure, particularly in internal medicine due to the high number of admissions from emergency departments, with a significant proportion of patients suffering from cardiac decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Sujet majeur (≥18 ans)
* Diagnostic d'amylose à TTR suite à une hospitalisation en médecine interne aux HUS entre 01/01/2013 au 31/12/2023.

Exclusion Criteria:

* Subject (and/or their legal representative, if applicable) who has expressed their opposition to the reuse of their data for scientific research purposes.
* Type of amyloidosis other than ATTR after review of the medical record (immunological assessment, imaging assessment, expert report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sujet majeur (≥18 ans) avec un diagnostic d'amylose à TTR
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Describe the number of cases of transthyretin (TTR) cardiac amyloidosis referred to internal medicine between 2013 and 2023. | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Interne - CHU de Strasbourg - France, Strasbourg, France